CLINICAL TRIAL: NCT06198361
Title: Value of Whole-body SPECT-CT CzT-based Camera (VERITON-CT) in the Assessment of Chronic Inflammatory Rheumatism With Axial Involvement (ASOCE)
Brief Title: Value of Whole-body SPECT-CT CzT-based Camera (VERITON-CT) in the Assessment of Chronic Inflammatory Rheumatism With Axial Involvement
Acronym: ASOCE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Isabelle Chary-Valckenaere, Head of Rhumatology, Central Hospital, Nancy, France
Other Study IDs: 2023PI091
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Spondyloarthritis
Keywords: spondyloarthritis; sacroiliitis; sacroiliac joints; VERITON-CT; SPECT-CT; thoracolumbar spine
MeSH Terms: conditions — Spondylarthritis; Sacroiliitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis of chronic inflammatory rheumatism with axial involvement is not always easy, and is fraught with difficulties : radiological sacroiliitis is not an early sign of spondyloarthritis and the delay in detecting radiological signs contributes to the delay in diagnosis.

Nevertheless, spondyloarthritis is now the second most common chronic inflammatory rheumatic disease, affecting 0.43% of the french population.

The aim of this retrospective study is to evaluate the diagnostic performance of whole-body SPECT-CT CzT-based camera (VERITON-CT) in the assessment of chronic inflammatory rheumatism with axial involvement

MRI of the sacroiliac joints and thoracolumbar spine were used as a gold standard.

DETAILED DESCRIPTION:
The present study was conducted by the Department of Rheumatology and Nuclear Medicine of the University Hospital Centre of Nancy (France).

An initial number of 51 hospitalised patients (35 females, 16 males) who underwent SPECT-CT CzT-based camera for polyarthralgia or spinal pain between November 2021 and February 2023 and initial suspicion of chronic inflammatory rheumatism were included in the study.

The investigators retrospectively reviewed the electronic medical records of the consecutive patients using medical softwares (DxCare or VNA Philips). The investigators collected demographic data (age, gender), clinical data (anamnesis, pain level (EVA) and location, standardized clinical activity scores like Ankylosing Spondylitis Disease Activity Score (ASDAS), Widespread Pain Index (WPI), symptom severity scale (SSS)), biological data (protein chain reaction in milligrams per litre), and medical imaging data (X-rays, MRI and CT scans).

The data collected was entered into an Excel spreadsheet protected by a security code.

For medical imaging data, the investigators performed a reading of the sacroiliac and thoracolumbar spine medical imaging under the supervision of an experienced rheumatologist specialising in chronic inflammatory rheumatism.

The investigators assessed the diagnostic performance of VERITON-CT (sensitivity, specificity), using MRI of the sacroiliac joints and thoracolumbar spine as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised patients (hospitalisation sector or day hospital)
* Patients who underwent SPECT-CT CzT-based camera for polyarthralgia or spinal pain between November 2021 and February 2023
* Patients who underwent axial MRI
* Initial suspicion of chronic inflammatory rheumatism

Exclusion Criteria:

* Patients who did not give their consent
* Patients with extravasation of contrast agent at the injection site
* Patients with a missing phase on SPECT-CT (Blood-Pool phase or Delayed phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 78 patients with SPECT-CT
  Among them : 51 patients with axial MRI (spine n=42 and/or sacroiliac joints n=47) :
  * 1 excluded for extravasation of contrast agent at the injection site
  * 1 excluded for "blood- pool phase" SPECT missing
  For a total of n = 47 patients (sacroiliac MRI); 25 classified as spondyloarthritis : axial spondyloarthritis, ankylosis spondylitis, psoriatic arthritis, SAPHO syndrome ; And 22 non-spondyloarthritis : Fibromyalgia, osteoarthritis, rheumatoid arthritis, Bertolotti syndrom, scoliosis, familial Mediterranean fever…
  For a total of n = 42 patients (thoracolumbar MRI); 22 patients in spondyloarthritis group (15 spondyloarthritis, 4 psoriatic arthritis and 3 SAPHO syndrome) and 20 in non-spondyloarthritis group (1 rheumatoid arthritis, 2 fibromyalgia, 13 osteoarthritis, 1 familial Mediterranean fever, 2 arthralgia in IBD and 1 arthralgia in cystic fibrosis).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
SI MRI (binary) | November 1, 2021 to February 1, 2023
  Positives MRI of the sacroiliac joints, according to the ASAS (Assessment of SpondyloArthritis international Society) criteria : binary value
MRI SPARCC (Spondyloarthritis Research Consortium of Canada) Score | November 1, 2021 to February 1, 2023
  SPARCC scores of the sacroiliac joints and of the thoracolumbar spine in MRI : quantitative value.
  Thoraco-lumbar SPARCC score : from 0 to 108, higher scores means worst outcome SI SPARCC score : from 0 to 72, higher scores means worst outcome
SI BP phase (binary) | November 1, 2021 to February 1, 2023
  Positives sacroiliac joints data in VERITON-CT (Blood-Pool phase) : binary value
SI D phase (binary) | November 1, 2021 to February 1, 2023
  Positives sacroiliac joints data in VERITON-CT (Delayed phase) : binary value
SI SUV (Standardized Uptake Values) BP phase | November 1, 2021 to February 1, 2023
  Sum of the SUVs of the sacroiliac joints measured on VERITON-CT (Blood-Pool Phase) : quantitative value
Thoracolumbar SUV (Standardized Uptake Values) BP phase | November 1, 2021 to February 1, 2023
  Sum of the SUVs of the thoracolumbar spine measured on VERITON-CT (Blood-Pool Phase) : quantitative value
SI SUV D phase | November 1, 2021 to February 1, 2023
  Sum of the SUVs of the sacroiliac joints measured on VERITON-CT (Delayed Phase) : quantitative value
Thoracolumbar SUV D phase | November 1, 2021 to February 1, 2023
  Sum of the SUVs of the thoracolumbar spine measured on VERITON-CT (Delayed Phase) : quantitative value
Thoracolumbar MRI (binary) | November 1, 2021 to February 1, 2023
  Positives MRI of the thoracolumbar spine, ≥3 inflammatory discovertebral corners : binary value
Thoracolumbar BP phase (binary) | November 1, 2021 to February 1, 2023
  Positives thoracolumbar spine data in VERITON-CT (Blood-Pool phase) : binary value
Thoracolumbar D phase (binary) | November 1, 2021 to February 1, 2023
  Positives thoracolumbar spine data in VERITON-CT (Delayed phase) : binary value

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MORIZOT, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costantino F, Talpin A, Said-Nahal R, Goldberg M, Henny J, Chiocchia G, Garchon HJ, Zins M, Breban M. Prevalence of spondyloarthritis in reference to HLA-B27 in the French population: results of the GAZEL cohort. Ann Rheum Dis. 2015 Apr;74(4):689-93. doi: 10.1136/annrheumdis-2013-204436. Epub 2013 Dec 18. PMID 24351517
- [Background] Pialat JB, Di Marco L, Feydy A, Peyron C, Porta B, Himpens PH, Ltaief-Boudrigua A, Aubry S. Sacroiliac joints imaging in axial spondyloarthritis. Diagn Interv Imaging. 2016 Jul-Aug;97(7-8):697-708. doi: 10.1016/j.diii.2016.02.013. Epub 2016 Mar 31. PMID 27050638
- [Background] Pipikos T, Kassimos D, Angelidis G, Koutsikos J. Bone Single Photon Emission/Computed Tomography in the Detection of Sacroiliitis in Seronegative Spondyloarthritis: A Comparison with Magnetic Resonance Imaging. Mol Imaging Radionucl Ther. 2017 Oct 3;26(3):101-109. doi: 10.4274/mirt.50570. PMID 28976332